CLINICAL TRIAL: NCT04540939
Title: Neural Mechanisms of Mindfulness-based Cognitive Therapy (MBCT) for Posttraumatic Stress Disorder (PTSD) - COVID Substudy
Brief Title: Neural Mechanisms of Mindfulness-based Cognitive Therapy (MBCT) for PTSD - COVID Related Substudy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Anthony P King, Associate Professor of Psychiatry and Behavioral Health, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00152509-COVID Substudy; 1R61AT009867 (NIH)
Record Dates: First submitted 2020-09-04; First posted 2020-09-07 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Trauma
Keywords: Mindfulness-Based Cognitive Therapy; Muscle Relaxation; Group Psychotherapy
MeSH Terms: conditions — Wounds and Injuries | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician will not know the group assignment until blind is broken. Statistician randomizes the groups. Principal investigator will not know group assignment until blind is broken.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): MBCT is a "mindfulness-based intervention" group intervention involving in session and at home practicve of mindfulness meditation and other mindfulness practices. There are8 sessions each with a specific theme and and these are ~2 hours long. Over the 8-weeks participants will learn several mindfulness meditation techniques. Each session will involve group discussion and feedback. Participants will be asked to practice these techniques at home, and keep a log of mood, and stress ratings.
  Audio files with exercises will be given to participants so that they can practice at home between sessions.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Muscle Relaxation Therapy (Active Comparator): PMR is a relaxation-based group intervention similar to other relaxation interventions commonly used for anxiety and PTSD. It involves in session and at home practicve of relaxation techniques including tensing and relaxing muscle groups, but no specifici mindfulness or meta-cogntive awaremess instructions. This PMR group has been designed as an active comparator with similar stucture to MBCT, but without mindfulness instruction. There are 8 sessions each with a specific theme and these are ~2 hours long. Over the 8-weeks participants will learn several relaxation techniques. Each session will involve group discussion and feedback. Participants will be asked to practice these techniques at home, and keep a log of mood, and stress ratings.
  Audio files with exercises will be given to participants so that they can practice at home between sessions.
  Interventions: Behavioral: Muscle Relaxation Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — There will be 8 sessions and these will be approximately 2 hours long. Over the 8-weeks participants will learn several mindfulness meditation techniques. Each session will involve group discussion and feedback. Participants will be asked to practice these techniques at home, and keep a log of mood, and stress ratings.
  Audio files with exercises will be given to participants so that they can practice at home between sessions.
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Behavioral: Muscle Relaxation Therapy — Each MR session is approximately 2 hours. Over the 8-weeks you will learn how to relax your body using a step-by-step process in which you alternate between squeezing and relaxing your muscles. You will learn about your body's natural response to stress and how to use muscle relaxation during your everyday life. Each session will also involve group discussion and feedback. You will be asked to practice these techniques at home, and keep a log of your mood, and stress ratings. You will receive audio files with exercises so you can practice at home between sessions.
  Arms: Muscle Relaxation Therapy

SUMMARY:
This clinical trial is a sub-study to treat participants that were not eligible in the main study (HUM00152509/NCT03874793) to receive MBCT or MRT in hard hit COVID-19 areas with trauma history and current COVID-related distress.

The purpose of this treatment-only sub-study is to see how eligible participants with life history of any trauma and are currently experiencing elevated COVID-related stress are affected by two different PTSD therapies involving Mind-Body practices; Mindfulness based Cognitive Therapy (MBCT) and Muscle Relaxation Therapy.

The targeted individuals will reside in areas (Washtenaw, Wayne, and Oakland counties in Michigan, etc.) that have been affected by COVID-19. Participants will have assessments before and after 8 weeks of therapy (remote MBCT or MRT).

DETAILED DESCRIPTION:
This clinical trial is a sub-study to treat participants that were not eligible in the main study (HUM00152509/NCT03874793) to receive MBCT or MRT in hard hit COVID-19 areas with trauma history and current COVID-related distress.

The purpose of this treatment-only sub-study is to see how eligible participants with life history of any trauma and are currently experiencing elevated COVID-related stress are affected by two different PTSD therapies involving Mind-Body practices; Mindfulness based Cognitive Therapy (MBCT) and Muscle Relaxation Therapy.

The targeted individuals will reside in areas (Washtenaw, Wayne, and Oakland counties in Michigan, etc.) that have been affected by COVID-19. Participants will have assessments before and after 8 weeks of therapy (remote MBCT or MRT).

ELIGIBILITY:
Inclusion Criteria:

* COVID distress sample: resides in geographical area heavily impacted by COVID-19 have a history of trauma
* Has current elevated levels of COVID related stress and/or distress (worry, repetitive negative thinking) (COVID stress scale score > 15, worry / repetitive negative thinking, Penn State Worry Questionnaire (PSWQ) score >35 ).

Exclusion Criteria:

* PTSD
* Suicide risk
* Psychosis
* Life history of schizophrenia
* Current substance dependence
* Other factors that preclude safe and meaningful participation in the study, at discretion of the PI and study team

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS-adult short form level 2) Anxiety survey | up to 8 weeks
  This Anxiety-Adult measure 7-item PROMIS Anxiety Short Form assesses the pure domain of anxiety in individuals age 18 and older. The participants will select how often they have been bothered by symptoms during the past 7 days from 1=never to 5=always (the higher the score the more anxiety).
Penn State Worry Questionnaire (PSWQ-16) Worry survey | up to 8 weeks
  The PSWQ is a well-validated self-administered, 16-item, Likert-type scale designed to measure worry. Possible range of scores is 16-80 with the algorithm of Total scores: 16-34 Low Worry, 35-59 Moderate, and 60-80 High Worry.
PROMIS (adult short form) Emotional Depression survey | up to 8 weeks
  This is an 8 question survey where participants will select answers of 1= Never to 5= always. The higher the score the greater severity of depression.
Working Alliance Inventory- short revised (WAI-SR) | up to 8 weeks
  This is a 12-item measure that assesses therapy clients' perception of working alliance with their therapists, developed by Adam Horvath with 3 factors of shared goals, tasks, and personal bond / regard. The participants select from Seldom= 1, Sometimes=2, Fairly often =3, Very often = 4, and Always = 5. The higher the score the higher working alliance.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS-adult short form level 2) Anxiety survey group differences (MBCT and PMR) | up to 8 weeks
  This Anxiety-Adult measure 7-item PROMIS Anxiety Short Form assesses the pure domain of anxiety in individuals age 18 and older. The participants will select how often they have been bothered by symptoms during the past 7 days from 1=never to 5=always (the higher the score the more anxiety). This will look at the group differences between MBCT and PMR.
Penn State Worry Questionnaire (PSWQ-16) Worry survey group differences (MBCT and PMR) | up to 8 weeks
  The PSWQ is a well-validated self-administered, 16-item, Likert-type scale designed to measure worry. Possible range of scores is 16-80 with the algorithm of Total scores: 16-34 Low Worry, 35-59 Moderate, and 60-80 High Worry. This will look at the group differences between MBCT and PMR.
PROMIS (adult short form) Emotional Depression survey group differences (MBCT and PMR) | up to 8 weeks
  This is an 8 question survey where participants will select answers of 1= Never to 5= always. The higher the score the greater severity of depression. This will look at the group differences between MBCT and PMR.
Working Alliance Inventory- short revised (WAI-SR) group differences (MBCT and PMR) | up to 8 weeks
  This is a 12-item measure that assesses therapy clients' perception of working alliance with their therapists, developed by Adam Horvath with 3 factors of shared goals, tasks, and personal bond / regard. The participants select from Seldom= 1, Sometimes=2, Fairly often =3, Very often = 4, and Always = 5. The higher the score the higher working alliance.This will look at the group differences between MBCT and PMR.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony King, Ph.D., Principal Investigator — University of Michigan; David Fresco, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
We plan to make available data from human subjects initially to collaborators for independent replication / data pooling. Completely de-identified research data (redacted according to NIH practice to prevent disclosure of personal identifiers) which documents the research findings will be made available after the main findings from the finalized research dataset have been accepted for publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 36 months of completion of the project.
Access Criteria: Access to data generated by the project will be available for educational, research and non-profit purposes to researchers who provide a methodologically sound proposal. Data generated under this project will be administered in accordance with NIH Sharing policies, including NIH Policy on Dissemination of NIH-Funded Clinical Trial Information (8/2016), and the NIH Grants Policy Statement (Availability of Research Results) (11/2015). Depending on such NIH policies, Data generated by this project may be available for educational, research or non-commercial purposes under the terms of a data use agreement. Data will be stored in an established data repository (e.g. Inter-university Consortium for Political and Social Research (ICPSR): icpsr.umich.edu) with appropriate provisions for curation and longterm preservation.